CLINICAL TRIAL: NCT03962764
Title: Growing Responsible Fathers Descriptive Program Evaluation
Status: Completed | Type: Observational
Sponsor: University of North Florida (Other)
Collaborators: Northeast Florida Healthy Start Coalition (Unknown)
Responsible Party: Principal Investigator, Jeff Will, Professor of Sociology, Director, NE FL Center for Community Initiatives, University of North Florida
Other Study IDs: 16-012
Record Dates: First submitted 2018-10-02; First posted 2019-05-24 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2020-03

CONDITIONS: Father-Child Relations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community: Community fathers include fathers who are recruited through community partners and self-referrals. Only fathers 18 years of age and older are included in program analysis
  Interventions: Behavioral: Responsible Fatherhood Program

INTERVENTIONS:
Behavioral: Responsible Fatherhood Program — 24 hours of fatherhood curriculum, 6 hours of financial literacy, workforce development, and case management.

SUMMARY:
The overall evaluation plan for the Growing Responsible Fathers program (Fatherhood PRIDE) will utilize both a process evaluation and an outcomes evaluation, and will include both quantitative and qualitative approaches. Pre- and post-test surveys will be used to measure short-term outcomes outlined in the logic model including whether or not there has been an increase in self-efficacy and knowledge related to personal finance, parent engagement, healthy relationships, and education. Pre-test surveys will be administered at intake and/or prior to program activity and post-test surveys will be conducted at the conclusion of the program activity.

DETAILED DESCRIPTION:
The overall evaluation plan for the Growing Responsible Fathers program (Fatherhood PRIDE) will utilize both a process evaluation and an outcomes evaluation, and will include both quantitative and qualitative approaches. Pre- and post-test surveys will be used to measure short-term outcomes outlined in the logic model including whether or not there has been an increase in self-efficacy and knowledge related to personal finance, parent engagement, healthy relationships, and education. Pre-test surveys will be administered at intake and/or prior to program activity and post-test surveys will be conducted at the conclusion of the program activity.

Intermediate outcomes will be measured using a follow-up survey at six (6) months after completing the primary components of the program. The follow-up surveys will be administered via a variety of methods in order to increase response rates and will measure outcomes identified in the logic model such as knowledge and self-efficacy.

Additional attempts will be made online through an email invitation as well as with phone calls. Center for Community Initiatives staff will be responsible for conducting the follow-up surveys with the program participants. Focus groups will be conducted with a volunteer sample of participants at the end of their program workshops to assess satisfaction with the program, what worked, and what could be improved.

ELIGIBILITY:
Inclusion Criteria:

* Fathers or father figure

Exclusion Criteria:

-

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males, identify male
Study Population: The program will serve 1350 fathers in Baker, Clay, Duval, Nassau and St. Johns' counties in the five year project period. Fathers are referred by the local family courts, re-entry centers and the federal and state Healthy Start programs; the child welfare system; and other community partners. The program serves two sub-populations: incarcerated fathers and community fathers.
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Increased knowledge gain | post test after 12 week program (incarcerated) or 4-6 weeks (community)
  Do participants who complete the program increase knowledge gains in financial literacy, co-parenting skills, and responsible fatherhood/family relationships after participating in program as measured by pre/post test. The outcome measure for each domain (financial literacy, co-parenting skills, and responsible fatherhood/family relationships) will be a total calculated from the number of correctly answered questions adapted from the curriculum.
Increased self-efficacy | Post test after 4-6 week program (community)
  Do Community participants who complete the program increase self-efficacy to pay for child support as measured by pre/post test. The outcome measure will be a total of six scores (range 0-100) to statements related to paying child support.
Increased engagement | Post test after 4-6 week program (community) and 6 month followup survey
  Do Community Participants who complete the program increase self reported engagement with their children as measured by pre/post test. The outcome measure will be a total of six scores (range 0-4) of various engagement activities with youngest child. These engagement measures were adapted from the FRPN Father Engagement Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Will, Principal Investigator — University of North Florida

IPD SHARING:
Plan to Share IPD: No